CLINICAL TRIAL: NCT02313129
Title: Causes of Comorbid Infertility Among Women With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00057614
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-04

CONDITIONS: Infertility; Rheumatoid Arthritis
Keywords: Infertility; Rheumatoid Arthritis
MeSH Terms: conditions — Infertility; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood tests
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Rheumatoid Arthritis: This group will complete questionnaires related to prior pregnancies, intentions and goals for childbearing, fertility history and detailed menstrual history. They will also have a physical exam and blood tests.
- Healthy Controls: This group will complete questionnaires related to prior pregnancies, intentions and goals for childbearing, fertility history detailed menstrual history, and blood tests.

SUMMARY:
The purpose of this study is to increase our understanding of infertility in women with Rheumatoid Arthritis (RA). In this study the study team will compare the differences in ovarian reserve (the ability to provide egg cells that are capable of fertilization), the frequency of ovulation and the number of pregnancies between women with and without RA. It is possible that RA activity and medications limit ovarian reserve and ovulation, which may increase infertility among women with RA. There are several suspected causes for infertility in RA, including age-related fertility decline, inflammatory changes that impact endometrial receptivity and discourage implantation, accelerated ovarian decline due to certain arthritis medications and increased frequency of anovulation (a menstrual cycle during which ovaries do not release an egg) due to RA activity.

This study is the first step toward our long term goal of increasing the ability of all women with RA to build the family they desire.

ELIGIBILITY:
Inclusion Criteria:

1. RA cohort: Women diagnosed with RA (2010 ACR/EULAR criteria) at least one year prior to enrollment
2. Healthy cohort: Women without autoimmune disease

Exclusion Criteria:

1. Unilateral or bilateral ovarian surgery
2. Prior exposure to known or possible ovary-toxic medications (e.g., cyclophosphamide, other chemotherapeutic agents)

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Rheumatoid Arthritis Women and Health Control Women
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-08; Primary Completion 2017-01-24 (Actual); Study Completion 2017-01-24 (Actual)

PRIMARY OUTCOMES:
Ovarian Reserve between women with and without RA | At study enrollment
Ovulation Frequency between women with and without RA | At study enrollment

SECONDARY OUTCOMES:
Rates of Infertility between women with and without RA | At study enrollment
Number of Pregnancies between women with and without RA | At study enrollment
Age at attempted and actual conception between women with and without RA | At study enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Megan Clowse, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States